CLINICAL TRIAL: NCT03781687
Title: Bilateral vs. Unilateral Erector Spinae Plane Block for Laparoscopic Cholecystectomy; A Randomised Controlled Trial
Brief Title: Bilateral vs. Unilateral Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Can AKSU, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: KIA 2018/488
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Pain; Cholecystitis; Gallstone
Keywords: erector spinae plane block; postoperative pain; laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative; Cholecystitis; Gallstones

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral (Active Comparator): Bilateral ESP block will be performed
  Interventions: Procedure: Bilateral ESP Block; Device: Intravenous Morphine patient controlled analgesia device
- Unilateral (Active Comparator): Unilateral ESP block will be performed
  Interventions: Procedure: Unilateral ESP Block; Device: Intravenous Morphine patient controlled analgesia device

INTERVENTIONS:
Procedure: Bilateral ESP Block — Bilateral ESP Block will be performed at T8
  Arms: Bilateral
Procedure: Unilateral ESP Block — Unilateral ESP Block will be performed at T8 (right side)
  Arms: Unilateral
Device: Intravenous Morphine patient controlled analgesia device — 24 hour morphine consumption will be recorded

SUMMARY:
The importance of multimodal analgesia for postoperative pain management is well known and regional anesthesia techniques are commonly prefferred to provide better analgesia. Erector spinae plane block (ESB) is a new defined and effective regional anesthesia technique. But two injections can be unconfortable for some patients. With this study, we aimed to compare the analgesia effect of bilateral and unilateral ESP block for laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Pateints undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* obesity (body mass index >35 kg/m2)
* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* coagulopathy
* recent use of analgesic drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | preoperative 24th hour
  Morphine consumption will be recorded

SECONDARY OUTCOMES:
Numeric Rating Scale | postoperative 24th hour
  A NRS involves asking the patient to rate his or her pain from 0 to 10 (11 point scale) with the understanding that 0 is equal to no pain and 10 is equal to worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Can Aksu, Principal Investigator — Kocaeli Üniversitesi Tıp Fakültesi
Locations (1):
- Kocaeli University Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No